CLINICAL TRIAL: NCT03033381
Title: A Comparison of Preoperative and Postoperative Testicular Volume and Blood Flow in Patients With Inguinal Hernia, Hydrocele, and Cord Cyst: A Prospective Cohort Study
Brief Title: A Comparison of Testicular Volume and Blood Flow in Patients With Inguinal Hernia, Hydrocele, and Cord Cyst
Acronym: IHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocatepe University (Other)
Responsible Party: Principal Investigator, Ahmet Ali Tuncer, Asst Prof Dr, Kocatepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-KAEK-86/05-80
Record Dates: First submitted 2017-01-05; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Inguinal Hernia Repair
Keywords: Children; Inguinal hernia; Testis; Doppler ultrasonography
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: operated and nonoperated side testis of each patient accepted two different group.
Who Masked: Outcomes Assessor
Masking Description: Statistician was masking
Oversight: Data Monitoring Committee: No

ARMS (2):
- operated side testis (Active Comparator): Operated side testis volume and blood flow will be evaluated with color doppler ultrasound before and after the surgery (Preoperative, 7 day and 30 day)
  Interventions: Device: Color Doppler Ultrasound
- Contralateral testis (Sham Comparator): Nonoperated side testis volume and blood flow will be evaluated with color doppler ultrasound before and after the surgery (Preoperative, 7 day and 30 day)
  Interventions: Device: Color Doppler Ultrasound

INTERVENTIONS:
Device: Color Doppler Ultrasound — Radiological evaluation was performed by a single radiologist using CDUS for operated side testis of each patient preoperatively and on days 7 and 30 post-surgery. Longitudinal, anteroposterior, and transverse diameters of the testis were measured, and the testicular volume was calculated automatically using the CDUS device (volume = 0.523 × D1 × D2 × D3, where D1, D2, and D3 were the maximal longitudinal, anteroposterior, and transverse diameters defined by CDUS) for both testicles in each patient . Peak systolic velocity (PSV) was calculated using the CDUS system (in cm3/s) for both testicles in each patient.
  Other Names: Operated side testis
  Arms: operated side testis
Device: Color Doppler Ultrasound — Radiological evaluation was performed by a single radiologist using CDUS for nonoperated side testis of each patient preoperatively and on days 7 and 30 post-surgery. Longitudinal, anteroposterior, and transverse diameters of the testis were measured, and the testicular volume was calculated automatically using the CDUS device (volume = 0.523 × D1 × D2 × D3, where D1, D2, and D3 were the maximal longitudinal, anteroposterior, and transverse diameters defined by CDUS) for both testicles in each patient . Peak systolic velocity (PSV) was calculated using the CDUS system (in cm3/s) for both testicles in each patient.
  Other Names: Nonoperated side testis
  Arms: Contralateral testis

SUMMARY:
Here, investigators aimed to evaluate the effect of inguinal operations performed with a modified Ferguson technique upon testicular volume and blood flow. This study involved 23 patients receiving surgery for inguinal hernia, hydrocele, and cord cyst. The color Doppler ultrasound (CDUS) was used to assess testicular volume and blood flow before and after a modified Ferguson technique surgery. The pre- and postoperative testicular volume and blood flow were compared with the contralateral testes. Statistical Package for the Social Sciences (SPSS) software was used to statistically analyze the data arising; the Mann-Whitney U test and Friedman test were used to compare samples, and P < 0.05 was accepted as statistically significant.

DETAILED DESCRIPTION:
Patients and Methods The study was performed prospectively with the approval of the Local Human Ethics Committee. All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards. All patients included in the study were provided with a patient consent form.

Study Group The analysis included male patients who were younger than 17 years and possessing one-sided inguinal hernia, hydrocele, or cord cyst and who were otherwise healthy. The study was performed prospectively between April 2016 and June 2016 in a medical faculty pediatric surgery unit.

Study plan Following diagnosis, patients received a CDUS and testicular volume and blood flow were measured preoperatively. All patients then received surgery with modified Ferguson repair. Testicular volume and blood flow were then reassessed by CDUS on days 7 and 30 following surgery.

Radiological evaluation Radiological evaluation was performed by a single radiologist using color doppler ultrasound (CDUS) preoperatively and on days 7 and 30 post-surgery. Longitudinal, anteroposterior, and transverse diameters of the testis were measured, and the testicular volume was calculated automatically using the CDUS device (volume = 0.523 × D1 × D2 × D3, where D1, D2, and D3 were the maximal longitudinal, anteroposterior, and transverse diameters defined by CDUS) for both testicles in each patient [1]. Peak systolic velocity (PSV) was calculated using the CDUS system (in cm3/s) for both testicles in each patient.

Statistical analysis The SPSS 15.0 (Statistical Package for the Social Sciences) software package was used for all statistical analysis. Testicular volumes and blood flow were analyzed as mean±standard deviation. The Mann-Whitney U test was used to compare differences in testicular volume and blood flow between the testis receiving surgery and the contralateral testis. Differences in preoperative, early postoperative (7 days post-surgery), and late postoperative (30 days post-surgery) testicular volume and blood flow of each testicle were compared using the Friedman test and P < 0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Our analysis included boys who were younger than 17 years and possessing one-sided inguinal hernia, hydrocele, or cord cyst and who were otherwise healthy.

Exclusion Criteria:

* Patients who had bilaterally inguinal hernia, hydrocele, or cord cyst

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change of testicular volume | Change of testicular volume from preoperative to postoperative 30 days
  Radiological evaluation was performed by a single radiologist using CDUS preoperatively and on days 7 and 30 post-surgery. Longitudinal, anteroposterior, and transverse diameters of the testis were measured, and the testicular volume was calculated automatically using the CDUS device (volume = 0.523 × D1 × D2 × D3, where D1, D2, and D3 were the maximal longitudinal, anteroposterior, and transverse diameters defined by CDUS) for both testicles in each patient
Change of blood flow | Change of blood flow from preoperative to postoperative 30 days
  Radiological evaluation was performed by a single radiologist using CDUS preoperatively and on days 7 and 30 post-surgery. Peak systolic velocity (PSV) was calculated using the CDUS system (in cm3/s) for both testicles in each patient.

IPD SHARING:
Plan to Share IPD: No